CLINICAL TRIAL: NCT02694978
Title: A Phase III, Randomized, Multicenter, Double-Blind, Safety Study of Ferumoxytol Compared to Ferric Carboxymaltose for the Treatment of Iron Deficiency Anemia (IDA)
Brief Title: A Phase III Safety Study of Ferumoxytol Compared to Ferric Carboxymaltose for the Treatment of Iron Deficiency Anemia (IDA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMAG-FER-IDA-304
Record Dates: First submitted 2016-02-08; First posted 2016-03-01 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency anemia; IDA; ferumoxytol; ferric carboxymaltose; FCM; Injectafer; Feraheme; Ferinject
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide; ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferumoxytol (Experimental): Participants received an IV infusion of ferumoxytol 510 milligram (mg) diluted (17 milliliter [mL]) in 233 mL 0.9% sodium chloride injection, United States Pharmacopeia (USP) (normal saline) (final volume 250 mL) over at least 15 minutes with a second dose 7-8 days after the first dose, for a total cumulative dose of 1.020 g.
  Interventions: Drug: Ferumoxytol
- FCM (Active Comparator): Participants received an IV infusion of FCM 750 mg diluted (15 mL) in 235 mL 0.9% sodium chloride injection, USP (normal saline) (final volume 250 mL) over at least 15 minutes with a second dose 7-8 days after the first dose, for a total cumulative dose of 1.500 g.
  Interventions: Drug: FCM

INTERVENTIONS:
Drug: Ferumoxytol
  Other Names: Feraheme
  Arms: Ferumoxytol
Drug: FCM
  Other Names: Injectafer, Ferinject
  Arms: FCM

SUMMARY:
To evaluate the safety of 1.020 grams (g) of intravenous (IV) ferumoxytol compared to 1.500 g of IV ferric carboxymaltose (FCM).

ELIGIBILITY:
Key Inclusion Criteria include:

* Participants with IDA and in whom IV iron treatment is indicated and defined as:

  * Participants with documented hemoglobin <12.0 g per deciliter (dL) for females and <14.0 g/dL for males within 60 days of dosing And
  * Participants with documented transferrin saturation (TSAT) ≤20% or Ferritin ≤100 nanograms (ng) per mL within 60 days of dosing
* Documented history of unsatisfactory oral iron therapy or in whom oral iron cannot be tolerated, or for whom oral iron is considered medically inappropriate (as per oral iron history questionnaire)
* All participants (male and female) of childbearing potential who are sexually active who agree to routinely use adequate contraception from randomization throughout the duration of the study

Key Exclusion Criteria include:

* Known hypersensitivity reaction to any component of ferumoxytol or FCM
* History of allergy to an IV iron
* History of multiple drug allergies
* Participants with dialysis-dependent chronic kidney disease
* Hemoglobin ≤7.0 g/dL
* Female participants who are pregnant, intend to become pregnant, are breastfeeding, have a positive serum/urine pregnancy test or not willing to use effective contraceptive precautions during the study (including females of childbearing potential who are partners of male participants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2014 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (108):
- United States (86):
  - Clinical Trial Site, Huntsville, Alabama
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Anaheim, California
  - Clinical Trial Site, Chula Vista, California
  - Clinical Trial Site, Corona, California
  - Clinical Trial Site, Encino, California
  - Clinical Trial Site, Fountain Valley, California
  - Clinical Trial Site, Granada Hills, California
  - Clinical Trial Site, La Mesa, California
  - Clinical Trial Site, Orange, California
  - Clinical Trial Site, Oxnard, California
  - Clinical Trial Site, Riverside, California
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, West Hollywood, California
  - Clinical Trial Site, Westminster, California
  - Clinical Trial Site, Bristol, Connecticut
  - Clinical Trial Site, Norwalk, Connecticut
  - Clinical Trial Site, Clearwater, Florida
  - Clinical Trial Site, Gainesville, Florida
  - Clinical Trial Site, Lauderdale Lakes, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Miami Lakes, Florida
  - Clinical Trial Site, North Miami, Florida
  - Clinical Trial Site, South Miami, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Winter Haven, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Augusta, Georgia
  - Clinical Trial Site, Savannah, Georgia
  - Clinical Trial Site, Thomasville, Georgia
  - Clinical Trial Site, Elk Grove Village, Illinois
  - Clinical Trial Site, Evergreen Park, Illinois
  - Clinical Trial Site, Hazel Crest, Illinois
  - Clinical Trial Site, Skokie, Illinois
  - Clinical Trial Site, Wichita, Kansas
  - Clinical Trial Site, Crestview Hills, Kentucky
  - Clinical Trial Site, Metairie, Louisiana
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Bethesda, Maryland
  - AMAG Pharmaceuticals, Inc., Waltham, Massachusetts
  - Clinical Trial Site, Bay City, Michigan
  - Clinical Trial Site, Flint, Michigan
  - Clinical Trial Site, Saginaw, Michigan
  - Clinical Trial Site, Chesterfield, Missouri
  - Clinical Trial Site, Kansas City, Missouri
  - Clinical Trial Site, Kirksville, Missouri
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, East Setauket, New York
  - Clinical Trial Site, Flushing, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Rosedale, New York
  - Clinical Trial Site, Asheville, North Carolina
  - Clinical Trial Site, Charlotte, North Carolina
  - Clinical Trial Site, Greensboro, North Carolina
  - Clinical Trial Site, Hickory, North Carolina
  - Clinical Trial Site, Jacksonville, North Carolina
  - Clinical Trial Site, Morehead City, North Carolina
  - Clinical Trial Site, Raleigh, North Carolina
  - Clinical Trial Site, Wilmington, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Marion, Ohio
  - Clinical Trial Site, Norman, Oklahoma
  - Clinical Trial Site, Tulsa, Oklahoma
  - Clinical Trial Site, Jenkintown, Pennsylvania
  - Clinical Trial Site, Levittown, Pennsylvania
  - Clinical Trial Site, Scottdale, Pennsylvania
  - Clinical Trial Site, Smithfield, Pennsylvania
  - Clinical Trial Site, Upland, Pennsylvania
  - Clinical Trial Site, Greenville, South Carolina
  - Clinical Trial Site, Greer, South Carolina
  - Clinical Trial Site, Rapid City, South Dakota
  - Clinical Trial Site, Germantown, Tennessee
  - Clinical Trial Site, Kingsport, Tennessee
  - Clinical Trial Site, Memphis, Tennessee
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, Fort Sam Houston, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Longview, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Schertz, Texas
  - Clinical Trial Site, Orem, Utah
  - Clinical Trial Site, Fredericksburg, Virginia
  - Clinical Trial Site, Norfolk, Virginia
  - Clinical Trial Site, Seattle, Washington
- Canada (3):
  - Clinical Trial Site, Sault Ste. Marie, Ontario
  - Clinical Trial Site, Vaughan, Ontario
  - Clinical Trial Site, Montreal, Quebec
- Hungary (5):
  - Clinical Trial Site, Budapest
  - Clinical Trial Site, Debrecen
  - Clinical Trial Site, Komárom
  - Clinical Trial Site, Szekszárd
  - Clinical Trial Site, Vác
- Latvia (5):
  - Clinical Trial Site, Jelgava
  - Clinical Trial Site, Krāslava
  - Clinical Trial Site, Liepāja
  - Clinical Trial Site, Riga
  - Clinical Trial Site, Ventspils
- Lithuania (5):
  - Clinical Trial Site, Kaunas
  - Clinical Trial Site, Klaipėda
  - Clinical Trial Site, Šiauliai
  - Clinical Trial Site, Utena
  - Clinical Trial Site, Vilnius
- Poland (3):
  - Clinical Trial Site, Bialystok
  - Clinical Trial Site, Warsaw
  - Clinical Trial Site, Wroclaw
- Clinical Trial Site, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adkinson NF, Strauss WE, Macdougall IC, Bernard KE, Auerbach M, Kaper RF, Chertow GM, Krop JS. Comparative safety of intravenous ferumoxytol versus ferric carboxymaltose in iron deficiency anemia: A randomized trial. Am J Hematol. 2018 May;93(5):683-690. doi: 10.1002/ajh.25060. Epub 2018 Feb 24. PMID 29417614
- [Background] Adkinson NF, Strauss WE, Bernard K, Kaper RF, Macdougall IC, Krop JS. Comparative safety of intravenous Ferumoxytol versus Ferric Carboxymaltose for the Treatment of Iron Deficiency Anemia: rationale and study design of a randomized double-blind study with a focus on acute hypersensitivity reactions. J Blood Med. 2017 Sep 26;8:155-163. doi: 10.2147/JBM.S142236. eCollection 2017. PMID 29033620
- [Derived] Wolf M, Chertow GM, Macdougall IC, Kaper R, Krop J, Strauss W. Randomized trial of intravenous iron-induced hypophosphatemia. JCI Insight. 2018 Dec 6;3(23):e124486. doi: 10.1172/jci.insight.124486. PMID 30518682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with iron deficiency anemia (IDA), <12.0 grams (g) per deciliter (dL) for females and <14.0 g/dL for males within 60 days of dosing and transferrin saturation (TSAT) <20% or Ferritin ≤100 nanograms (ng) per milliliter (mL) within 60 days of dosing and a history of unsatisfactory oral iron therapy or in whom oral iron could not be used.
Groups:
- Ferric Carboxymaltose (FCM): Participants received an IV infusion of FCM 750 mg diluted (15 mL) in 235 mL 0.9% sodium chloride injection, USP (normal saline) (final volume 250 mL) over at least 15 minutes with a second dose 7-8 days after the first dose, for a total cumulative dose of 1.500 g.
Period: Overall Study
Arm/Group | Ferumoxytol | Ferric Carboxymaltose (FCM)
Started | 1006 | 1008
Received at Least 1 Dose of Study Drug | 997 | 1000
Completed (Completed=received at least 1 dose of study drug and returned for final study visit (Week 5).) | 935 | 948
Not Completed | 71 | 60
Not completed — Adverse Event | 10 | 9
Not completed — Withdrawal by Subject | 22 | 19
Not completed — Lost to Follow-up | 14 | 17
Not completed — Death | 4 | 1
Not completed — Other-Decision of Participant | 6 | 1
Not completed — Other-Investigator's decision | 1 | 0
Not completed — Other-Unable to be reached | 0 | 1
Not completed — Other-Protocol noncompliant | 2 | 1
Not completed — Other-Personal reasons | 3 | 3
Not completed — Other-Withdrew prior to dosing | 9 | 8

BASELINE CHARACTERISTICS:
Population: The safety population included any randomized participant who received any amount of study drug. Treatment group was based on actual treatment.
Groups:
- Ferumoxytol: Participants received an IV infusion of ferumoxytol 510 mg diluted (17 mL) in 233 mL 0.9% sodium chloride injection, USP (normal saline) (final volume 250 mL) over at least 15 minutes with a second dose 7-8 days after the first dose, for a total cumulative dose of 1.020 g.
- Total: Total of all reporting groups
Arm/Group | Ferumoxytol | Ferric Carboxymaltose (FCM) | Total
Number analyzed (Participants) | 997 | 1000 | 1997
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (17.30) | 54.8 (17.02) | 55.2 (17.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 743 | 776 | 1519
  Male | 254 | 224 | 478

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent (TE) Moderate To Severe Hypersensitivity Reactions (Rxns), Including Anaphylaxis, Or Moderate To Severe Hypotension
Description: All IV iron formulations carry some risk of serious hypersensitivity reactions or anaphylaxis. Signs and symptoms potentially representing hypersensitivity were recorded and adjudicated by a blinded Clinical Events Committee (CEC). Hypotension is defined as a >30% drop in systolic blood pressure from baseline or decrease of >20 mmHg for systolic blood pressure.
  Statistical analysis was only performed on composite data. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after first dosing) through Week 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ferumoxytol | Ferric Carboxymaltose (FCM)
Number analyzed (Participants) | 997 | 1000
Participants
  Moderate hypersensitivity reaction | 3 | 6
  Severe hypersensitivity reaction | 1 | 0
  Anaphylaxis | 0 | 0
  Moderate hypotension | 2 | 1
  Severe hypotension | 0 | 0
  Any TE moderate to severe hypersensitivity rxn | 6 | 7
Statistical Analysis 1: Comparison: Ferumoxytol vs Ferric Carboxymaltose (FCM); Statistical analysis was only performed on composite reaction data (that is, the "Any TE moderate to severe hypersensitivity rxn" row in the data table); Test type: Non-Inferiority — The non-inferiority margin of 2.64% was used for the primary endpoint statistical analysis; p = 0.0001, Wald; The p-value was calculated using the Wald large sample assumption; Treatment difference = -0.10, 95% CI 2-sided [-0.80 to 0.61]

2. Secondary Outcome: Participants With Moderate To Severe Hypersensitivity Reactions, Including Anaphylaxis, Serious Cardiovascular Events, And Death
Description: All IV iron formulations carry some risk of serious hypersensitivity reactions or anaphylaxis. Signs and symptoms potentially representing hypersensitivity were recorded and adjudicated by a blinded Clinical Events Committee (CEC).
  A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after first dosing) through Week 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ferumoxytol | Ferric Carboxymaltose (FCM)
Number analyzed (Participants) | 997 | 1000
Participants
  Moderate hypersensitivity reaction | 3 | 6
  Severe hypersensitivity reaction | 1 | 0
  Anaphylaxis | 0 | 0
  Serious cardiovascular event | 6 | 13
  Death | 4 | 2
  Any moderate to severe hypersensitivity rxn | 13 | 20

3. Secondary Outcome: Mean Change In Hemoglobin From Baseline To Week 5
Description: Mean change in hemoglobin from Baseline to Week 5 was calculated for each participant as: Hemoglobin Change = Hemoglobin (Week 5) - Hemoglobin (Baseline). Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information.
Time Frame: Baseline (Day 1), Week 5
Population: Intent-to-treat (ITT) population: any randomized participant who had any exposure to study drug, based on randomized treatment assignment.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferumoxytol | Ferric Carboxymaltose (FCM)
Number analyzed (Participants) | 997 | 1000
g/dL | 1.38 (1.351) | 1.63 (1.535)

4. Secondary Outcome: Mean Change In Hemoglobin Per Gram Of Iron Administered From Baseline To Week 5
Description: Mean change in hemoglobin per g of iron administered from Baseline (Day 1) to Week 5 was calculated for each participant as: Hemoglobin Change = Hemoglobin (Week 5) - Hemoglobin (Baseline). Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information.
Time Frame: Baseline (Day 1), Week 5
Population: ITT population: any randomized participant who had any exposure to study drug, based on randomized treatment assignment.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferumoxytol | Ferric Carboxymaltose (FCM)
Number analyzed (Participants) | 997 | 1000
g/dL | 1.35 (1.353) | 1.10 (1.050)

ADVERSE EVENTS:
Arm/Group | Ferumoxytol | Ferric Carboxymaltose (FCM)
Serious Adverse Events (participants affected / at risk) | 36/997 | 35/1000
Other Adverse Events (participants affected / at risk) | 186/997 | 245/1000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ferumoxytol (N=997) | Ferric Carboxymaltose (FCM) (N=1000)
Seizure (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 3 | 3
Gastroenteritis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Cardiorespiratory arrest (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Joint abscess (Infections and infestations) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/743 | 0/776
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/743 | 0/776
Completed suicide (Psychiatric disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Post-procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/743 | 1/776
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferumoxytol (N=997) | Ferric Carboxymaltose (FCM) (N=1000)
Nausea (Gastrointestinal disorders) | 35 | 60
Diarrhoea (Gastrointestinal disorders) | 29 | 33
Abdominal pain (Gastrointestinal disorders) | 17 | 21
Constipation (Gastrointestinal disorders) | 14 | 13
Vomiting (Gastrointestinal disorders) | 11 | 13
Fatigue (General disorders) | 30 | 36
Chest discomfort (General disorders) | 8 | 11
Pyrexia (General disorders) | 7 | 22
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 12
Headache (Nervous system disorders) | 60 | 82
Dizziness (Nervous system disorders) | 25 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 11
Flushing (Vascular disorders) | 11 | 16
Hypertension (Vascular disorders) | 7 | 15
Chest pain (General disorders) | 10 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data have been received by Sponsor, the Site, and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 180 days to allow Sponsor to protect its interests.